CLINICAL TRIAL: NCT03933293
Title: A Phase 2 Study to Evaluate the Safety and Efficacy of PCSK9 Inhibitor AK102 in Patients With Homozygous Familial Hypercholesterolemia (HoFH)
Brief Title: A Study to Evaluate the Safety and Efficacy of the PCSK9 Inhibitor AK102 in Patients With HoFH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akeso (Industry)
Collaborators: AD Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK102-202
Record Dates: First submitted 2019-04-28; First posted 2019-05-01 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Homozygous Familial Hypercholesterolemia
Keywords: HoFH; LDL-C
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK102 (Experimental): 450mg AK102, Q4W, subcutaneous injection
  Interventions: Drug: AK102; Drug: Statins; Drug: Ezetimibe
- placebo (Placebo Comparator): Placebo, Q4W, subcutaneous injection
  Interventions: Drug: Statins; Drug: Ezetimibe

INTERVENTIONS:
Drug: AK102 — 450mg, Q4W, subcutaneous injection
  Arms: AK102
Drug: Statins — Lipid-lowering therapies
Drug: Ezetimibe — Lipid-lowering therapies

SUMMARY:
AK102 is being developed for the treatment of HoFH. The study will be conducted in 2 parts, part 1 is open label, single arm study to evaluate the safety, tolerability and efficacy of PCSK9 inhibitor AK102, and part 2 is double blind, randomized, placebo controlled study to evaluate the efficacy and safety of PCSK9 inhibitor AK102. The treatment period will last 12 week.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ≥18 years of age with a diagnosis of homozygous familial hypercholesterolemia by genetic confirmation or a clinical diagnosis based on a history of an untreated low-density lipoprotein cholesterol (LDL-C) concentration >500 mg/deciliter (dL) [13 millimoles/liter (mmol/L)] together with either xanthoma before 10 years of age or evidence of heterozygous familial hypercholesterolemia in both parents
* Stable on pre-existing, lipid-lowering therapies (statins in combination with ezetimibe) for at least 4 weeks with no planned medication or dose change for the duration of study participation
* Fasting central lab LDL-C concentration >130 mg/dL (3.4 mmol/L) and triglyceride concentration <400 mg/dL (4.5 mmol/L).
* Body weight of 40 kilograms (kg) or greater at screening

Exclusion Criteria:

* Received LDL plasma replacement therapy within 8 weeks before Investigational product administration
* Received Lomitapide or Mipomersen within 5 months before Investigational product administration
* Received prior treatment with PCSK9 inhibitors or AK102.
* Unexplained creatine kinase (CK) ≥ 5 times the upper limit of normal (ULN)
* Subjects with untreated chronic hepatitis B or chronic hepatitis B virus (HBV) DNA exceeding 500 IU/ mL or active hepatitis C virus (HCV) should be excluded. Subjects with non-active HBsAg carriers, treated and stable hepatitis B (HBV DNA <500 IU/ mL) , and cured hepatitis C can be enrolled. Subjects with positive HCV antibodies are eligible only if the HCV RNA test results are negative.
* Known allergic reactions to any ingredients of AK102
* Any other condition(s) that would compromise the safety of the patient or compromise the quality of the clinical study as judged by the Investigator and/or Medical Monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Percent Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Week 12 | Week 12
Incidence of treatment-emergent adverse events as assessed by CTCAE V5.0（only for part 1） | From baseline through 12 weeks

SECONDARY OUTCOMES:
Percent Change From Baseline in High-density lipoprotein (HDL) cholesterol | From baseline through 12 weeks
Percent Change From Baseline in non High-density lipoprotein (non-HDL) cholesterol | From baseline through 12 weeks
Percent Change From Baseline in Serum Triglyceride (TG) | From baseline through 12 weeks
Percent Change From Baseline in Apolipoprotein B (Apo B) | From baseline through 12 weeks
Percent Change From Baseline in Apolipoprotein A-I (Apo A-I) | From baseline through 12 weeks
Percent Change From Baseline in Total Cholesterol(TC) | From baseline through 12 weeks
Change From Baseline in Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) | From baseline through 12 weeks
Concentrations of AK102 in Serum | Part 1: Day 1,Day 2, Day 4, Day 8, Day 15, Day 22, D29, D57. Part 2: Day 1, Day 29, Day 57
Number of subjects who develop detectable anti-drug antibodies (ADAs) | From baseline through 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shuyang Zhang, MD, Principal Investigator — Peking Union Medical College Hospital; Lvya Wang, Principal Investigator — Beijing Anzhen Hospital
Locations (2):
- China (2):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No